CLINICAL TRIAL: NCT02117700
Title: Effect of N-acetyl Cysteine on Non Alcoholic Fatty Liver Disease in Obese Children
Brief Title: Fatty Liver Disease in Obese Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Babu Balagopal, Head, Obesity & Cardiovascular Research Laboratory, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NemoursCC; American Diabetes Association (Other Grant/Funding Number: ADA1-14-CE-04)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Nonalcoholic Fatty Liver Disease; Cardiovascular Disease
Keywords: fatty liver; obesity; children; oxidative stress; antioxidants
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Fatty Liver | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled randomized double blind
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N-acetyl cysteine-1 (Experimental): N-acetyl cysteine 600 mg once/day + Placebo once/day for 16 weeks
  Interventions: Dietary Supplement: N-acetyl cysteine 600 mg once/day
- N-acetyl cysteine-2 (Experimental): N-acetyl cysteine 600 mg twice/day for 16 weeks
  Interventions: Dietary Supplement: N-acetyl cysteine 600mg twice/day
- Placebo (Placebo Comparator): Placebo twice/day for 16 weeks
  Interventions: Other: Placebo twice/day

INTERVENTIONS:
Dietary Supplement: N-acetyl cysteine 600 mg once/day — NAC 600 mg once/day + Placebo once/day for 16 weeks
  Arms: N-acetyl cysteine-1
Dietary Supplement: N-acetyl cysteine 600mg twice/day — N-acetyl cysteine 600 mg twice/day for 16 weeks
  Arms: N-acetyl cysteine-2
Other: Placebo twice/day — Placebo capsules twice/day for 16 weeks
  Arms: Placebo

SUMMARY:
Although weight reduction through physical activity-based interventions is the mainstay therapy for nonalcoholic fatty liver disease (NAFLD), its maintenance is difficult and typically unsuccessful. This affirms the extreme need for alternate and/or adjunct therapies. Although convincing data from animal studies and a few adult human studies on the benefits of a natural product, N-acetyl cysteine (NAC), in a variety of liver conditions including NAFLD have emerged, studies in children are scarce. Therefore, the aim of the study is to test the use NAC as an innovative approach to attenuate the progression of NAFD in obese children with biopsy proven NASH. The central hypothesis is that NAC supplementation will reduce liver fat and liver enzymes and ameliorate risk factors of cardiometabolic disease in children with NAFLD.

DETAILED DESCRIPTION:
Physical activity (PA)-induced weight reduction, the suggested therapy for noalcoholic liver disease (NAFLD), is difficult and its maintenance is typically unsuccessful in children, affirming the acute need for alternative/adjunct therapies. Although few promising approaches have been reported, the benefits are incongruent and mostly marginal. N-acetyl cysteine (NAC), a derivative of the natural amino acid, cysteine, appears to be promising as an adjunct therapy to PA. Animal and a few adult human studies suggest NAC-induced attenuation of liver abnormalities, oxidative stress, insulin resistance and inflammation. The primary aim of the proposal is to determine in obese children with biopsy proven NASH and elevated liver enzymes the effect of NAC at two different doses on liver fat using magnetic resonance imaging (MRI), liver enzymes and risk factors of cardiometabolic disease. We hypothesize that NAC will produce beneficial effect on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years and older
* NASH confirmed in a previous biopsy
* HbAIc <6.4%
* ALT > 60 U/L or 1.5 times the upper limit of normal

Exclusion Criteria:

* Chronic liver disease including alpha-1-antitrypsin deficiency, Wilson's disease, autoimmune and viral hepatitis
* Medications such as adrenergic β-blockers, steroids and other drugs known to interfere with the measurement of liver enzymes and risk factors for cardiovascular disease
* Heart disease, chronic renal disease, adrenal, hepatic or thyroid dysfunction; active malignancy; and anemia
* History of prior treatment with NAC
* Evidence of hypersensitivity/allergy to NAC
* Alcoholism or drug abuse and smoking
* Inter-current illness over 7 days before the study & surgery in the past 3 mo.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in liver fat (MRI) and ALT levels from baseline and at 16 weeks | Upto 16 weeks
  The primary outcome will be sustained reduction in ALT level, defined as 50% or less of the baseline level or 40 U/L or less and significant changes in liver fat (MRI) at the end of the study. All measurements of biological factors will be performed in the post absorptive (fasted) state.

OTHER OUTCOMES:
Change in Biomarkers of cardiovascular disease from baseline and at 16 weeks | Upto 16 weeks
  The secondary outcome will be attenuation of abnormal levels of biomarkers of cardiovascular disease such as markers of inflammation, oxidative stress and insulin resistance. All measurements of biological factors will be performed in the post absorptive (fasted) state.

CONTACTS AND LOCATIONS:
Overall Officials: Babu Balagopal, PhD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic/Alfred I duPont Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No